CLINICAL TRIAL: NCT03444597
Title: Post-Market Clinical-Follow-Up Study of Suprasorb® C Collagen Wound Dressing
Acronym: Suprasorb®C
Status: Completed | Type: Observational
Sponsor: Lohmann & Rauscher (Industry)
Responsible Party: Sponsor
Other Study IDs: 2017-A02514-49
Record Dates: First submitted 2018-02-08; First posted 2018-02-23 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Venous or Mixed Leg Ulcers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Post-Market Clinical-Follow-Up Study of Suprasorb® C collagen wound dressing

DETAILED DESCRIPTION:
Prospective, uncontrolled multi-center, observational cohort study. The objectives of the PMCF study are confirmation of the performance, and to collect additional safety data regarding expected adverse events and to detect potential unexpected adverse events associated with use of Suprasorb®C under the conditions of routine use.

Suprasorb® C collagen wound dressing is a certified medical device (manufacturer: Lohmann & Rauscher International GmbH & Co. KG). The product has been marketed in the EU since 1983 as Opragen® (medicinal product), since 1995 as the medical device Opraskin® and since 2001 under the name Suprasorb C (medical device).

Suprasorb® C is intended to be used as a wound dressing for the support of wound healing or wound area reduction.

Participating Centers: 40 study nurses will participate to the PMCF Study Duration: 24 months Cohort size: 110 patients Follow-up: 8 weeks

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age and under 85 years of age
* Patient suffering from confirmed venous or mixed vascular leg ulcers
* Stagnating wound conditions, i.e. exudation phase > 2 months, not responding to traditional dressing and standard treatment (standard treatment is a clear definition and for venous ulcers compression should be included)
* Target ulcers between 2 cm and 10 cm in the largest diameter
* Written confirmation from the study nurse that the patient was informed, orally agreed to participate and to comply with study treatment and planned visits

Exclusion Criteria:

Use of Suprasorb® C collagen wound dressing is contraindicated according to the current IFU:

* Clinically infected areas
* Presence of known allergies to one or several of its components.

In addition following patients shall not be included into this study:

* Patient not covered by health insurance/social security
* Patient suffering serious life threatening disease
* Pregnant or breastfeeding women
* Minor patient, protected adult, person without liberty

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient population is patient with venous or mixed leg ulcers
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2018-01-24 (Actual); Primary Completion 2020-01-23 (Actual); Study Completion 2020-01-23 (Actual)

PRIMARY OUTCOMES:
Progression of healing after application of Suprasorb® C collagen wound dressing is used as parameter for performance evaluation | Progression of healing is assessed at 8 weeks
  Progression of healing after application of Suprasorb® C collagen

SECONDARY OUTCOMES:
Frequency and severity of adverse events | Frequency and severity is assessed up to 8 weeks
  Frequency and severity of adverse events, incidences, as well as known risk and side effects, i.e. wound infection, side effects in the group of allergic disorders, pain, and maceration

CONTACTS AND LOCATIONS:
Overall Officials: Daria TROFIMENKO, Study Director — Lohmann and Rauscher
Locations (1):
- RCTs, Lyon, France